CLINICAL TRIAL: NCT00704457
Title: Impact Of Sacral Neuromodulation On Urine Markers For IC
Brief Title: Impact Of Sacral Neuromodulation On Urine Markers For Interstitial Cystitis (IC)
Status: Completed | Type: Observational
Sponsor: Kenneth Peters, MD (Other)
Collaborators: Corewell Health East (Other)
Responsible Party: Sponsor-Investigator, Kenneth Peters, MD, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Other Study IDs: 2004-024
Record Dates: First submitted 2008-06-24; First posted 2008-06-25 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Interstitial Cystitis
Keywords: Interstitial Cystitis; IC; Sacral Nerve Stimulation
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urines were collected and sent for urine marker analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: One arm study. Urine collection.

SUMMARY:
Urine will be collected and sent to the University of Maryland. Urines will be analyzed for urine markers.

DETAILED DESCRIPTION:
Urine will be collected and flash frozen in liquid nitrogen then placed in a -70 C freezer. All urine will be collected and stored until the final follow-up is complete. The urine samples will then be sent as a single batch to the Department of Infectious Disease, University of Maryland. Urines will be assayed in a blinded fashion and a written report of the levels of each of the 3 urine markers will be sent to Beaumont Hospital. Change in urine marker levels will be analyzed and correlated with change in symptom scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be drawn from Dr. Peters patient base that covers Southeast Michigan.

Exclusion Criteria:

* Male

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone sacral nerve stimulation.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2004-02; Primary Completion 2006-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The purpose of this study is measure urine biomarkers levels in patients with interstitial cystitis who have elected to undergo sacral nerve stimulation as a treatment modality for their disease. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, MD, Principal Investigator — Corewell Health East
Locations (1):
- Beaumont Hospital - Royal Oak, Royal Oak, Michigan, United States